CLINICAL TRIAL: NCT01685892
Title: A Phase Ib Multicenter Dose-Finding and Safety Study of Venetoclax and Obinutuzumab in Patients With Relapsed or Refractory or Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study of Venetoclax in Combination With Obinutuzumab in Participants With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GP28331; 2012-002038-34 (EudraCT Number); NCT02339181 (obsolete NCT alias)
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose-Finding: Schedule A: Relapsed/Refractory CLL (Experimental): All 4 cohorts will begin venetoclax administration after the ramp-up period of 5 weeks. In 4 cohorts of participants with relapsed/refractory CLL escalating doses of venetoclax will be administered in combination with fixed dose obinutuzumab in the dose-finding stage. In Schedule A, venetoclax will be introduced before obinutuzumab. Schedule A will be explored prior to Schedule B.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Dose-Finding: Schedule B: Relapsed/Refractory CLL (Experimental): In 4 cohorts of participants with relapsed/refractory CLL escalating doses of venetoclax will be administered in combination with fixed dose obinutuzumab in the dose-finding stage. In Schedule B, venetoclax will be introduced after obinutuzumab. Schedule A will be explored prior to Schedule B.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Dose-Finding: Schedule A: Previously Untreated CLL (Experimental): All 4 cohorts will begin venetoclax administration after the ramp-up period of 5 weeks. In 4 cohorts of participants with previously untreated CLL escalating doses of venetoclax will be administered in combination with fixed dose obinutuzumab in the dose-finding stage. In Schedule A, venetoclax will be introduced before obinutuzumab. Schedule A will be explored prior to Schedule B.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Dose-Finding: Schedule B: Previously Untreated CLL (Experimental): In 4 cohorts of participants with previously untreated CLL escalating doses of venetoclax will be administered in combination with fixed dose obinutuzumab in the dose-finding stage. In Schedule B, venetoclax will be introduced after obinutuzumab. Schedule A will be explored prior to Schedule B.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Safety Expansion: Relapsed/Refractory CLL (Experimental): In participants with relapsed/refractory CLL a recommended dose of venetoclax will be administered in combination with obinutuzumab in the safety expansion stage. Schedule A or B will be used for the expansion cohort after a review of available safety data from the dose finding stage.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- Safety Expansion: Previously Untreated CLL (Experimental): In participants with previously untreated CLL a recommended dose of venetoclax will be administered in combination with obinutuzumab in the safety expansion stage. Schedule A or B will be used for the expansion cohort after a review of available safety data from the dose finding stage.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive IV infusion of obinutuzumab 100 milligrams (mg) on Day 1 of Cycle 1, 900 mg on Day 2 of Cycle 1, and 1000 mg on Days 8 and 15 of Cycle 1 and on Day 1 of Cycles 2-6.
  Other Names: GA101; RO5072759
Drug: Venetoclax — Participants will receive multiple doses of venetoclax orally once daily.
  Other Names: ABT-199, GDC-0199

SUMMARY:
This multi-center, open-label, dose-finding study will evaluate the safety and pharmacokinetics as well as the preliminary efficacy of venetoclax (GDC-0199; ABT-199) administered in combination with obinutuzumab to participants with relapsed/refractory or previously untreated chronic lymphocytic leukemia (CLL). The study is comprised of two stages for each participant population: a dose-finding stage and a safety-expansion stage. The dose-finding stage will explore multiple doses of venetoclax to be used in combination with a fixed dose of obinutuzumab. The dose-finding stage will also explore two schedules for drug administration, Schedule A (venetoclax introduced before obinutuzumab) and Schedule B (venetoclax introduced after obinutuzumab).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing/refractory or previously untreated chronic lymphocytic leukemia
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to (</=) 1
* Adequate bone marrow function
* Adequate coagulation, renal and hepatic function
* For all participants, agreement to remain abstinent or use contraceptive methods that result in a failure rate of less than (<) 1% per year during the treatment period and for at least 90 days (30 days for women) after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer

Exclusion Criteria:

* Participants who have undergone allogenic stem cell transplant are ineligible unless they meet the following criteria, a) participants who are off all immunosuppressive therapy, b) participants who have no signs and/or symptoms of acute or chronic graft versus host disease, or c) participants must have appropriate hematology counts
* Infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Investigational or anti-cancer therapy within 5 half-lives prior to the first dose of study drug
* History of significant renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities (DLTs) | Schedule (Sch) A (Cycle 1 Day 1 to Day 21), Sch B (Cycle 1 Day 22 to Cycle 2 Day 28) (1 Cycle=28 days)
Maximum Tolerated Dose (MTD) of Venetoclax in Combination with Obinutuzumab | Sch A (Cycle 1 Day 1 to Day 21), Sch B (Cycle 1 Day 22 to Cycle 2 Day 28) (1 Cycle=28 days)

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to end of study (up to approximately 5 years and 5 months)
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) to Obinutuzumab | Baseline up to Cycle 6 (1 Cycle=28 days)
Area Under the Concentration-Time Curve (AUC) of Venetoclax | Baseline up to Cycle 6 (1 Cycle=28 days)
Time to Maximum Observed Plasma Concentration (Tmax) of Venetoclax | Baseline up to Cycle 6 (1 Cycle=28 days)
Maximal Plasma Concentration (Cmax) of Venetoclax | Baseline up to Cycle 6 (1 Cycle=28 days)
Minimum Plasma Concentration (Cmin) of Venetoclax | Baseline up to Cycle 6 (1 Cycle=28 days)
Cmax of Obinutuzumab | Baseline up to Cycle 6 (1 Cycle=28 days)
Cmin of Obinutuzumab | Baseline up to Cycle 6 (1 Cycle=28 days)
Percentage of Participants with Confirmed Complete Response (CR) as Determined by Standard CLL Response Criteria | Baseline up to end of study (up to approximately 5 years and 5 months)
Percentage of Participants with Objective Response (Partial Response [PR] or CR [Including Cytopenic CR] as Determined by Standard CLL Response Criteria | Baseline up to end of study (up to approximately 5 years and 5 months)
Duration of Objective Response as Determined by Standard CLL Response Criteria | Baseline up to end of study (up to approximately 5 years and 5 months)
Overall Survival | Baseline up to death or end of study (up to approximately 5 years and 5 months)
Progression-Free Survival as Determined by Standard CLL Response Criteria | Baseline up to end of study (up to approximately 5 years and 5 months)
Change from Baseline in Number of B-Cells | Baseline up to end of study (up to approximately 5 years and 5 months)
Change from Baseline in Number of T-Cells | Baseline up to end of study (up to approximately 5 years and 5 months)
Change from Baseline in Number of Natural Killer (NK) Cells | Baseline up to end of study (up to approximately 5 years and 5 months)
Change from Baseline in Serum Immunoglobulin Level | Baseline up to end of study (up to approximately 5 years and 5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (10):
- United States (7):
  - UCSD Moores Cancer Center, La Jolla, California
  - Colorado Blood Cancer Institute (CBCI) at Presbyterian/ St. Luke's Medical Center, Denver, Colorado
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oncology Associates of Oregon, Springfield, Oregon
  - SCRI-Tennessee Oncology, Nashville, Tennessee
  - The Methodist Hospital Research Institute; Academic Office of Clinical Trials, Houston, Texas
- United Kingdom (3):
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary NHS Trust, Leicester
  - Barts and The London School of Medicine and Dentistry; Queen Mary, University of London, London

REFERENCES:
- [Derived] Samineni D, Gibiansky L, Wang B, Vadhavkar S, Rajwanshi R, Tandon M, Sinha A, Al-Sawaf O, Fischer K, Hallek M, Salem AH, Li C, Miles D. Pharmacokinetics and Exposure-Response Analysis of Venetoclax + Obinutuzumab in Chronic Lymphocytic Leukemia: Phase 1b Study and Phase 3 CLL14 Trial. Adv Ther. 2022 Aug;39(8):3635-3653. doi: 10.1007/s12325-022-02170-w. Epub 2022 Jun 16. PMID 35708885
- [Derived] Flinn IW, Gribben JG, Dyer MJS, Wierda W, Maris MB, Furman RR, Hillmen P, Rogers KA, Iyer SP, Quillet-Mary A, Ysebaert L, Walter HS, Verdugo M, Klein C, Huang H, Jiang Y, Lozanski G, Pignataro DS, Humphrey K, Mobasher M, Kipps TJ. Phase 1b study of venetoclax-obinutuzumab in previously untreated and relapsed/refractory chronic lymphocytic leukemia. Blood. 2019 Jun 27;133(26):2765-2775. doi: 10.1182/blood-2019-01-896290. Epub 2019 Mar 12. PMID 30862645